CLINICAL TRIAL: NCT03093454
Title: Effects of Lavender Oil on Postoperative Pain, Sleep Quality and Mood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scott Hollenbeck, MD (Other)
Collaborators: dōTERRA International (Industry)
Responsible Party: Sponsor-Investigator, Scott Hollenbeck, MD, Surgeon, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00071214
Record Dates: First submitted 2017-03-10; First posted 2017-03-28 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: Randomized study with control group and test group. Using a 1:1 treatment allocation ratio, the total of 60 patients (30 per arm) will be randomly assigned to control or treatment arm. The Statistical Investigator will generate the randomization scheme and monitor the randomization process over the course of the trial. The study will use randomization with random permuted blocks. The test group will receive 50% lavender oil diluted in fractionated coconut oil and the control group will have the current standard of care with no essential oil intervention. Fractionated coconut oil is being used because it is colorless, odorless, does not stain clothing, and has a long shelf life. It also serves as a carrier oil for the essential oil to absorb into the skin instead of evaporating off the skin due to essential oils volatile nature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention patient will receive current standard of care treatment and will answer surveys to collect data.
- Lavender Group (Experimental): Patient will receive lavender essential oil topically and by inhalation during their hospital stay while at the same time receiving regular standard of care.
  Interventions: Drug: Lavender Essential Oil

INTERVENTIONS:
Drug: Lavender Essential Oil — Lavender essential oil will be applied topically and by inhalation to the lavender group.
  Other Names: Lavandula angustifolia
  Arms: Lavender Group

SUMMARY:
This project will evaluate the integration of lavender essential oil in surgical patients during the perioperative and postoperative phase of care. The study will assess patients' pain, sleep quality, and mood. The goal is to support that lavender oil will decrease pain scores and narcotic use, increase sleep quality, and decrease anxiety by improving overall patient satisfaction and supporting their natural sense of well being. This research project will help support the use of complementary medicine in a hospital setting. The increased awareness and use of complementary medicine in a hospital setting will strengthen the patient centered care model that all hospitals strive to achieve.

DETAILED DESCRIPTION:
Background & Significance:

Essential oils have been formally documented in use since the time of the Egyptians. The Ebers Papyrus document notes Egyptians using frankincense for different physical ailments. In Greece Hippocrates used essential oils to fumigate the city of Athens to fight off the plague. In medieval periods lavender essential oil was used for its antidepressive, anxiolytic, sedative, and analgesic properties. Medieval Persian physicians made records of their treatment plans which included lavender for depression and pain for headaches. With the invention of steam distillation to separate the essential oil from the plant Europe began to use oils in perfumes and for medicinal benefits in the 1500's. Two physicians named Hieronymus and Brunschwig wrote one of the earliest printed books on the distillation and use of essential oils for medical benefits. By the 19th century a French chemist Rene- Maurice Gattefosse was known for studying essential oils and their therapeutic benefits. His work and documentation led the way for the support of essential oil in medical ailments. Robert Tisserand in the early 1990s reviewed the French chemists work and added to his research to help make essential oils more known to the public in present day.

In recent years lavender has been studied on human subjects to tests its known reputation for sedative, anxiolytic, and analgesic properties. In one clinical trial oral administration of lavender was compared to Ativan 0.5mg for generalized anxiety disorder. The study supported that the oral lavender oil called Silexan was as effective as 0.5mg of Ativan in adults with generalized anxiety disorder. A second clinical trial analyzing sleep quality found that ischemic heart patients in the intensive care unit received better sleep with 100% lavender oil undiluted placed on a cotton ball within 20cm from the patient from the hours of 9pm-6am. Two studies have used lavender oil through inhalation in the recovery room with an oxygen mask after surgery for pain control. The first study was patients after breast biopsy, the second was patients who just had laparoscopic adjustable gastric banding. The study with the breast biopsy patients showed a higher satisfaction rate with pain. The patients undergoing laparoscopic banding also showed a higher rate of satisfaction with pain as well as decreased opioid use in the recovery room. Furthermore one study used 100% lavender oil undiluted on the skin of pediatric patients undergoing tonsillectomy as a topical application and asked the patients to inhale. The study showed a decrease use in Tylenol usage postoperatively.

Design & Procedures:

Design Randomized study with control group and test group. Using a 1:1 treatment allocation ratio, the total of 60 patients (30 per arm) will be randomly assigned to control or treatment arm. The Statistical Investigator will generate the randomization scheme and monitor the randomization process over the course of the trial. The study will use randomization with random permuted blocks. The test group will receive 50% lavender oil diluted in fractionated coconut oil and the control group will have the current standard of care with no essential oil intervention. Fractionated coconut oil is being used because it is colorless, odorless, does not stain clothing, and has a long shelf life. It also serves as a carrier oil for the essential oil to absorb into the skin instead of evaporating off the skin due to essential oils volatile nature.

Study Procedure The lavender essential oil used will be from the company doTERRA. This essential oil company was chosen because this company has a medical and science governing board made up of physicians, surgeons, chemists and pharmacists. The oil is also third party tested by Dr. Robert Pappas a trusted chemist in the essential oil community for purity and quality. Gas chromatography and mass spectrometry are used to ensure purity and no unwanted substances are in the essential oil. doTERRA's essential oils have also already been used in a hospital setting at Vanderbilt University hospital in Tennessee. doTERRA's essential oils were diffused in the Vanderbilt ER at the nursing stations. After 3 months of diffusing staff felt less work related stress, less time feeling overwhelmed, and had more energy at work.

Study Interventions:

After informed consent is obtained, exactly 4 drops of 50% lavender solution will be placed on the wrist over the radial artery. The patient will rub her wrists and hands together and then inhale and exhale slowly for one minute. This will occur thirty minutes before being taken to the operating room. The dilution of 50% was chosen after reviewing Robert Tisserand's book on essential oil safety, consulting a local certified aromatherapist, Cynthia Loving, and consulting Dr. David Hill, executive vice president and chief medical officer of doTERRA essential oils. This percent dilution is recommended on skin and is not likely to cause irritation to the skin. Repeated insult patch skin testing from doTERRA has supported this dilution rate to be safe to the skin. Furthermore a previous study used 100 % lavender oil on children age 5-12 undergoing tonsillectomy with no adverse reactions. The first dose will be given thirty minutes prior to the operating room because it takes 20 minutes for lavender to be absorbed thought the skin and reach peak plasma levels.

During surgery the patient will receive 4 drops of 50% solution lavender oil on the temple region over the temporal artery every 2 hours until completion of surgery. This will be applied by the anesthesia team. If the temporal region is not accessible the shoulders or feet will be alternate locations of application. When the patient arrives to the recovery room she will receive lavender oil through an oxygen mask. A 50 % solution will be used by placing 4 drops of the lavender solution on the mask and wiping it around the mask with a cotton ball. This delivery method will be used because this was used in a study from New York University Medical Center studying postoperative pain and no adverse events occurred. When the patient is on the post-operative floor she will receive 50 % lavender oil on the wrist every 4 hours in the same manner as preoperatively from the hours of 6am to 9pm. Nightly (9pm-6am), 8 drops of 50% lavender oil will be placed on the cotton ball situated within 20cm of the patient. This method and concentration was chosen after reviewing a study in ischemic heart patients in the intensive care unit. The patients received lavender at bedside on a cotton ball and had statistically significant better sleep quality. The control group will have the current standard of care with no lavender intervention.

Blood pressure, pulse, respiratory rate, and oxygen saturation will be monitored in the preoperative area before lavender is given and 30 minutes after it is given. The level of pain will also be asked prior to application and at the second set of vitals. The control group will get two sets of vital measurements and pain scale measurements without any intervention.

The same vitals will be recorded while the patient is under anesthesia every 30 minutes. There will be a notation in the chart when lavender is given to correlate time from application to time of vitals recorded. A review of the electronic medical record will be done to record amount of narcotic needed interop in both groups.

In the recovery room after the patient is given lavender through the oxygen mask the same vital signs and pain score measurement will be taken 15, 30, and 60 minutes from lavender application. In the control group on arrival to the recovery room the same data points will be measured with the same time intervals with no intervention. The amount of narcotic needed in the recovery room will be taken from the electronic medical record for each group.

Postoperatively on the floor vital signs as noted above will be recorded every 4 hours. At each 4 hour interval after the vital signs are taken lavender will be applied to the experimental group and no intervention in the control group. One more set of vitals signs will be recorded 45min after application of lavender each time lavender is applied. There will be a review of narcotic use from the electronic medical record from both groups. There will be a notation when lavender was given to correlate lavender application and narcotic use.

The anxiety questionnaire will be given preop before the application of lavender and then daily for every post-op day they stay. The questionnaire is called the hospital anxiety and depression scale.

The sleep questionnaire will be given in preop before application of lavender and then daily for every post-op day they stay. The sleep questionnaire is called the Richard Campbell Sleep Questionnaire.

Daily starting on postop day 1 the patient will also record their level of satisfaction of pain control from a scale of 1-10 with 1 being not satisfied and 10 being satisfied. Patients typically stay in hospital 1-3 days post-op. A survey will be filled out daily.

Data Analysis & Statistical Considerations:

Study Design/Endpoints: The primary outcome will be a difference in pain scores between the 2 groups and/or decrease in narcotic use and/or increased patient satisfaction of pain control.

Secondary outcomes are better sleep and decreased anxiety. The secondary outcome will be a difference in scores from the two surveys, the Richards Campbell sleep questionnaire and the Hospital Anxiety Depression Scale.

Analytic Plan and Method: Differences in the change scores of pain in the two groups as well any other demographic and clinical continuous variables will be examined using t-test or Wilcoxon test, depending on whether the variables are normally or non-normally distributed respectively. The differences between the categorical variables will be examined using chi-squared or Fisher's exact test. Analysis will be conducted under the intention to treat (ITT). Missing data will be imputed under multiple imputation methods. Differences in the outcomes while controlling for potential covariates (age, etc) will be examined using linear regression. Significance of the tests will be assessed at alpha = 0.05. Analysis will be conducted using SAS 9.4 (SAS Institute, Inc., Cary, NC.).

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing any form of breast reconstruction therapy
* Ages 18-85
* At least a one night stay in hospital after surgery

Exclusion Criteria:

* Use of sleeping aide drugs
* Use of benzodiazepines
* History of any of the following: asthma, eczema, allergy to flowers, smell disorders
* Sensitivity to lavender oil or any of its ingredients
* Pregnant women will be excluded from the study. During routine preoperative testing the patient's menstrual history or urine pregnancy test will be performed to identify any patient who is pregnant.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hollenbeck, MD, Principal Investigator — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vakili N, Gorji A. Psychiatry and psychology in medieval Persia. J Clin Psychiatry. 2006 Dec;67(12):1862-9. doi: 10.4088/jcp.v67n1205. PMID 17194263
- [Background] Gorji A, Khaleghi Ghadiri M. History of headache in medieval Persian medicine. Lancet Neurol. 2002 Dec;1(8):510-5. doi: 10.1016/s1474-4422(02)00226-0. PMID 12849336
- [Background] Woelk H, Schlafke S. A multi-center, double-blind, randomised study of the Lavender oil preparation Silexan in comparison to Lorazepam for generalized anxiety disorder. Phytomedicine. 2010 Feb;17(2):94-9. doi: 10.1016/j.phymed.2009.10.006. Epub 2009 Dec 3. PMID 19962288
- [Background] Moeini M, Khadibi M, Bekhradi R, Mahmoudian SA, Nazari F. Effect of aromatherapy on the quality of sleep in ischemic heart disease patients hospitalized in intensive care units of heart hospitals of the Isfahan University of Medical Sciences. Iran J Nurs Midwifery Res. 2010 Fall;15(4):234-9. PMID 22049287
- [Background] Kim JT, Wajda M, Cuff G, Serota D, Schlame M, Axelrod DM, Guth AA, Bekker AY. Evaluation of aromatherapy in treating postoperative pain: pilot study. Pain Pract. 2006 Dec;6(4):273-7. doi: 10.1111/j.1533-2500.2006.00095.x. PMID 17129308
- [Background] Kim JT, Ren CJ, Fielding GA, Pitti A, Kasumi T, Wajda M, Lebovits A, Bekker A. Treatment with lavender aromatherapy in the post-anesthesia care unit reduces opioid requirements of morbidly obese patients undergoing laparoscopic adjustable gastric banding. Obes Surg. 2007 Jul;17(7):920-5. doi: 10.1007/s11695-007-9170-7. PMID 17894152
- [Background] Soltani R, Soheilipour S, Hajhashemi V, Asghari G, Bagheri M, Molavi M. Evaluation of the effect of aromatherapy with lavender essential oil on post-tonsillectomy pain in pediatric patients: a randomized controlled trial. Int J Pediatr Otorhinolaryngol. 2013 Sep;77(9):1579-81. doi: 10.1016/j.ijporl.2013.07.014. Epub 2013 Aug 8. PMID 23932834
- [Background] Koulivand PH, Khaleghi Ghadiri M, Gorji A. Lavender and the nervous system. Evid Based Complement Alternat Med. 2013;2013:681304. doi: 10.1155/2013/681304. Epub 2013 Mar 14. PMID 23573142
- [Background] Heidari Gorji MA, Ashrastaghi OG, Habibi V, Charati JY, Ebrahimzadeh MA, Ayasi M. The effectiveness of lavender essence on strernotomy related pain intensity after coronary artery bypass grafting. Adv Biomed Res. 2015 Jun 4;4:127. doi: 10.4103/2277-9175.158050. eCollection 2015. PMID 26261829

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Patient received coconut essential oil topically and by inhalation during their hospital stay while at the same time receiving regular standard of care.
  Coconut Essential Oil: will be applied topically and by inhalation to the control group.
  Completed daily surveys during inpatient stay in the hospital.
- Lavender Group: Patient received lavender essential oil topically and by inhalation during their hospital stay while at the same time receiving regular standard of care.
  Lavender Essential Oil: Lavender essential oil was applied topically and by inhalation to the lavender group.
  Completed daily surveys during inpatient stay in the hospital.
Period: Overall Study
Arm/Group | Control Group | Lavender Group
Started | 28 | 30
Completed | 22 | 27
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Scheduling conflict | 3 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Placebo/Control: Patient will receive coconut essential oil topically and by inhalation during their hospital stay while at the same time receiving regular standard of care.
  Coconut Essential Oil: Coconut essential oil will be applied topically and by inhalation to the control group.
- Total: Total of all reporting groups
Arm/Group | Placebo/Control | Lavender Group | Total
Number analyzed (Participants) | 22 | 27 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 26 | 45
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 26 | 47
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 13 | 20 | 33
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: Effects of Lavender Oil on Postoperative Pain Through Pain Scores
Description: Assess pain through pain scores documented in medical record compared to control group.
  Pain score of 0 is no pain versus pain score of 10 is highest pain possible.
Time Frame: Pre-operatively, Post-op Day 1 (POD1), and final post-op day (final POD)
Population: A total of 9 subjects were with drawn from the analysis as described in participant flow section. 58 subjects originally signed consent and 49 completed the study and used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Lavender Group
Number analyzed (Participants) | 22 | 27
score on a scale
  Preoperative | 0.5 (1.36) | 0.9 (1.80)
  Post-op Day 1 (POD1) | 3.5 (1.91) | 3.1 (2.74)
  Final Post-op Day (final POD) | 2.5 (1.92) | 2.9 (2.81)
Statistical Analysis 1: Comparison: Control Group vs Lavender Group; Lavender group compared to control group; Test type: Equivalence — Linear mixed effects models were used to investigate HADS scores (total, anxiety, and depression), sleep scores, and pain scores. Variables for time point (preoperative/Post-op Day 1/final Post-op Day) & arm were analyzed. Adjustment for multiple pairwise comparisons used the Scheffe method. Analyses were conducted based on the intent to treat principle. P-values<0.05 were considered statistically significant. Each time point, the mean and corresponding 95% confidence interval has been plotted; p = 0.05, Fisher Exact — The p value is calculated and adjusted for multiple comparisons; Odds Ratio (OR) = 95, Standard Deviation 1

2. Primary Outcome: Effects of Lavender Oil on Sleep
Description: Assess sleep quality by Richards Campbell sleep questionnaire survey A score of zero (0) minimal if any sleep at all versus 10 deep and sound sleeping during hospital stay.
Time Frame: Pre-operatively, Post-op Day 1(POD1), and final Post-op Day (final POD)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Lavender Group
Number analyzed (Participants) | 22 | 27
score on a scale
  Pre-operative | 6.5 (2.61) | 5.6 (2.39)
  Post-op Day 1 (POD1) | 5.5 (1.97) | 5.1 (2.08)
  Final Post-op Day (Final POD) | 6.6 (2.43) | 7.4 (1.71)

3. Primary Outcome: Effects of Lavender Oil on Mood
Description: Assess anxiety by hospital anxiety depression scale survey
  This 14-component scoring system is used to tabulate a total sum score (0-42) or separate anxiety and depression scores (0-21). A higher score represents a more severe degree of anxiety and/or depression. The severity of a patient's anxiety or depression may then be grouped into three categories based on the score (Normal, 0-7; Borderline abnormal, 8-10; Abnormal 11-21).
Time Frame: Pre-operatively, Post-op Day 1 (POD1), Final Post-op Day (Final POD)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Lavender Group
Number analyzed (Participants) | 22 | 27
units on a scale
  Pre-operative | 14.9 (1.68) | 14.4 (1.77)
  Post-op Day 1 (POD1) | 14.8 (2.14) | 15.0 (2.84)
  Final Post-op Day (Final POD) | 15.8 (2.77) | 15.7 (1.11)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout each patient's hospital stay during the time of essential oil application. Typically the AEs were collected over a 1 week period specifically when the essential oils were used. After each subject was discharged the study agent was no longer applied.
Description: No adverse events were to be found throughout the study.
Groups:
- Control: Patient will receive coconut essential oil topically and by inhalation during their hospital stay while at the same time receiving regular standard of care.
  Coconut Essential Oil: Coconut essential oil will be applied topically and by inhalation to the control group.
Arm/Group | Control | Lavender Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03093454/Prot_SAP_000.pdf